CLINICAL TRIAL: NCT06202482
Title: Enhance Physical Activity and Intergenerational Relationship Via Connect Active Program (CAP): a Pilot Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, TSE Mun Yee Mimi, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CAP
Record Dates: First submitted 2024-01-01; First posted 2024-01-11 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Elderly; Physical Inactivity
Keywords: Connective Active Program
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Participants in the intervention group will participate in a 6-week Connect Active Program (CAP). Young participants will be the pioneers and take the initiative to change their inactive and sedentary lifestyles by including exercise into their daily routines about once a week, at least 45 minutes each time. For instance, they could organize family field trips to waterfront parks or involve their older family members in their favorite sports. All walking activities included in the study should be done with the Nike Run Club App for record and outcome measures. For other activities in CAP, participants will use other apps following that week's topic. For instance, they will use Google Maps to search for the best routes to their destinations; transportation apps such as Kowloon Motor Bus, Long Win Bus, and Mass Transit Railway apps to search for stops and exits.
  Interventions: Other: Connect Active Program
- Control group (No Intervention): Participants in the control group will be provided with a leaflet as usual care. The pamphlet contains information about the benefits and some instructions for walking exercises for older adults.

INTERVENTIONS:
Other: Connect Active Program — Younger adults will help older adults increase their digital literacy, skills, and desire to exercise and become more physically active via the proposed intervention. The Connect Active Program will consist of two components: walking exercises and mobile apps.
  Arms: Experimental group

SUMMARY:
This study investigates how walking exercises and technology could enhance the quality of life in the older generation. It has three objectives: 1) To examine the effectiveness of the Connect Active Program (CAP) in improving intergenerational relationships, psychological well-being, and physical fitness for older adults; 2) To teach older adults to use mobile apps; 3) To examine the experiences and feedback from participants in using the apps and joining the CAP. This research will provide long-term insights into improving the overall health outcomes of older adults via intergenerational support and increasing the acceptance of mobile technology among older adults.

ELIGIBILITY:
Inclusion Criteria:

* Younger Adults/Participants:

  * Aged 18 to 30
  * Related to the older adult participant (i.e. family member, relatives)
  * Able to understand Cantonese
  * Own a smartphone and have access to the Internet
  * Able to take part in walking exercise and stretching program
* Older Adults/Participants:

  * Aged 60 or above
  * Able to understand Cantonese
  * Own a smartphone and have access to the Internet
  * Capable to participate in walking exercise and stretching program

Exclusion Criteria:

* Older Adults/Participants and Younger Adults/Participants:

  * Diagnosed with a mental disorder by neurologists or psychiatrists
  * With a history of drug addiction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
Aerobic Capacity and Endurance Evaluation with 6-Minute Walk Test (6MWT) | Baseline, Week 6
  It is initially created to assist in the examination of cardiopulmonary patients developed by the American Thoracic Society. It is a light-intensity exercise test to evaluate the aerobic capacity, endurance and oxygen saturation.

SECONDARY OUTCOMES:
Mobility and Balance Assessment with Time Up and Go Test | Baseline, Week 6
  To assess mobility, movement, static balance and dynamic in people with musculoskeletal impairments, conditions related to aging, quality of life, and pain. The instructions are given as standing up from a chair, walking 3 meters, turning, and back to sit.
Quality of Life Measurement | Baseline, Week 6
  Quality of life will be evaluated utilizing the World Health Organization Quality of Life-BREF (WHOQOL-BREF). It contains four realms: physical health, psychological health, social relationships, and environment. A 5-point response scale is used in the scale. WHOQOL-BREF has good validity and reliability.
Happiness Level Determination | Baseline, Week 6
  A 29-item measure of happiness; from 1 "strongly agree," to 6, "strongly disagree." The scale's reliability was 0.91.
Intergenerational Relationship Appraisal | Baseline, Week 6
  The intergenerational relationship quality scale (IRQS) to appraise the changes in intergenerational relationships, this questionnaire will allow the older participants to self-rate the relationship between the two generations. A 5-point response scale is applied in the scale.
Subjective Quality Assessment of Mobile Apps | Baseline, Week 6
  The 4-item subjective quality subscale of the Mobile Application Rating Scale (MARS) will be deployed to assess the overall quality of mobile apps involved in this study. MARS incorporates four objective quality subscales (engagement, functionality, aesthetics, and information quality) and one subjective quality subscale. Since a lengthy questionnaire would be complicated for the older participants to complete, we will only adopt the subjective quality subscale. All four items are assessed on a 5-point scale. The subjective quality subscale showed excellent internal consistency (alpha = 0.93) and interrater reliability intraclass correlation coefficient (ICC = 0.83). Higher scores indicate a higher level of subjective quality.
Participant Feedback Collection | Baseline, Week 6
  Semi-structured interview for older and younger participants: Individual interviews will be carried out by the Research Assistant upon completion of the CAP (post-test). They will be asked to comment on the perceived benefits, limitations and barriers in the program and the mobile apps, usefulness of the mobile apps, and recommendations for improving the CAP to meet their needs. Details of the questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Mimi MY Tse, PhD, Principal Investigator — School of Nursing and Health Studies, Hong Kong Metropolitan University
Locations (1):
- Hong Kong Metropolitan University, Kowloon, Hong Kong